CLINICAL TRIAL: NCT06133283
Title: High Intensity Endurance Exercise as a Primer to Virtual Reality for Optimizing Cortical Excitability and Neuroplasticity in Parkinson's Disease (PD)
Brief Title: Endurance Exercise & Virtual Reality for Optimizing Cortical Excitability and Neuroplasticity in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Anjali Sivaramakrishnan, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20230433H; 1K12TR004529-01 (NIH)
Record Dates: First submitted 2023-11-07; First posted 2023-11-15 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Aerobic exercise; Virtual reality; Rehabilitation; Balance; Neurophysiology
MeSH Terms: conditions — Parkinson Disease | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study will utilize a randomized controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity endurance exercise and virtual reality (experimental) (Experimental): The exercise group will perform high intensity interval exercise and VR-based games 3 times a week for 8 weeks.
  Interventions: Behavioral: High intensity endurance exercise; Behavioral: Virtual reality (VR)-based gaming
- Stretching and virtual reality (control) (Other): The stretching group will perform stretching exercises and VR-based games 3 times a week for 8 weeks.
  Interventions: Behavioral: Stretching exercise; Behavioral: Virtual reality (VR)-based gaming

INTERVENTIONS:
Behavioral: High intensity endurance exercise — High intensity interval exercise on a recumbent stepper for 30 minutes, 3 days per week.
  Arms: High intensity endurance exercise and virtual reality (experimental)
Behavioral: Stretching exercise — Stretches of face, neck, upper extremity, trunk and lower extremity muscles including whole body stretches for 30 minutes, 3 days per week.
  Arms: Stretching and virtual reality (control)
Behavioral: Virtual reality (VR)-based gaming — VR games will involve games that challenge balance such as reaching different targets during activities such as sit to stand, dodging obstacles etc. Participants will play approximately 6 games for 30 minutes, 3 days a week.

SUMMARY:
This study aims to determine the effects of aerobic exercise as a primer to add-on virtual reality (VR)-based rehabilitation on balance, postural control and neuroplasticity (ability of brain to adapt in structure and function) in individuals with Parkinson's disease (PD). This study will utilize two groups - one group will receive the exercise and VR, while the other group will receive stretching exercise and VR over eight weeks. The study team will administer outcomes at baseline, post-intervention (8 weeks) and follow-up (6 weeks after post-assessment).

DETAILED DESCRIPTION:
This study will enroll individuals diagnosed with Parkinson's disease who will be randomly assigned to 2 groups: 1) high intensity endurance exercise and virtual reality (experimental) or 2) stretching and virtual reality (control) for eight weeks (three sessions, thrice weekly). Outcomes will include balance and gait measures, blood-based biomarkers, neuroplasticity measures (assessed by transcranial magnetic stimulation), spinal reflex excitability (measured by H reflex) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD (ages 18 -85) in Hoehn and Yahr stages 2 - 3.
2. Subjects need to demonstrate a score of equal to or greater than 23 on the Mini Mental State Examination.
3. Subjects who have a score of ≤21.5 on the Mini Balance Evaluations Systems Test (miniBESTest).

Exclusion Criteria:

1. Subjects with a history of other neurological diseases (i.e., stroke, multiple sclerosis).
2. Subjects with a history of severe cardiopulmonary disease, uncontrolled hypertension, orthostatic hypotension, uncontrolled diabetes, severe osteoporosis, severe arthritis affecting their lower extremity joints.
3. Subjects with a history of PD-specific surgical procedures such as deep brain stimulation etc.
4. Subjects with a history of head injury.
5. Subjects with a history of seizures or epilepsy.
6. Subjects who are currently pregnant.
7. Individuals who use of medications that could alter corticomotor excitability or increase risk of seizure.
8. Individuals with skull abnormalities, fractures or unexplained, recurring headaches.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline, post (8 week), follow-up (14 weeks)
  Balance will be tested with the Mini Balance Evaluation Systems Test(miniBESTest), involving 14 different tasks including the timed up and go test to assess static and dynamic balance. Scores range from 0 to 28 with higher scores suggesting better balance.

SECONDARY OUTCOMES:
Postural stability | Baseline, post (8 week), follow-up (14 weeks)
  Postural stability will be assessed by the Biodex Balance System.
Endurance | Baseline, post (8 week), follow-up (14 weeks)
  The 6-minute walk test will be used as a measure of cardiovascular endurance
Spatiotemporal gait parameters | Baseline, post (8 week), follow-up (14 weeks)
  Spatiotemporal measures of gait will be acquired with the GAITRite™ gait mat.
Brain derived neurotrophic growth factor (BDNF) | Baseline, post (8 week), follow-up (14 weeks)
  Blood sample will be obtained for measuring circulating levels of brain derived neurotrophic growth factor (BDNF).
Corticomotor excitability | Baseline, post (8 week), follow-up (14 weeks)
  Corticomotor excitability for the tibialis anterior motor representations will be measured with single and paired pulse transcranial magnetic stimulation (TMS).
Spinal reflex excitability | Baseline, post (8 week), follow-up (14 weeks)
  H reflexes will be recorded for quantifying spinal reflex excitability. The H wave amplitude will be expressed as a % of the M wave amplitude (H/M ratio).
Parkinson's Disease Questionnaire (PDQ-39) | Baseline, post (8 week), follow-up (14 weeks)
  The Parkinson's disease questionnaire (PDQ-39) is a self report questionnaire that will be used to evaluate quality of life. The questionnaire consists of 39 items with each item being rated on a 5-point scale. Lower scores suggest higher quality of life.
Parkinson's Disease Cognitive Rating Scale (PD-CRS) | Baseline, post (8 week), follow-up (14 weeks)
  The Parkinson's disease cognitive rating scale will be used to test frontal subcortical tasks such as attention, working memory, verbal fluency and posterior cortical tasks such as confrontation naming and copying a clock. Scores range from 0 - 134 and higher scores suggest better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Sivaramakrishnan, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health San Antonio- Dept. of Physical Therapy, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected deidentified individual participant data (IPD) will be shared on an open source platform and summary results will be shared on ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication of the study findings.